CLINICAL TRIAL: NCT02941393
Title: Influence of Measurement Method of Labor Contractions on Labor Outcome and Newborn
Brief Title: Internal Versus External Tocodynamometry and Labor Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Central Finland Hospital District (Other)
Responsible Party: Principal Investigator, Tuija Hautakangas, Medical doctor, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R12229
Record Dates: First submitted 2016-09-07; First posted 2016-10-21 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Dystocia; Contractions
Keywords: internal tocodynamometry, external tocodynamometry, cesarean section, labor, newborn, vacuum extraction, dystocia
MeSH Terms: conditions — Dystocia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intrauterine pressure catheter (Active Comparator): Intrauterine pressure catheter is used during labor to follow up the contractions
  Interventions: Device: Intrauterine pressure catheter
- External tocodynamometry (Active Comparator): External tocodynamometry is used during labor to follow up the contractions
  Interventions: Device: External tocodynamometry

INTERVENTIONS:
Device: Intrauterine pressure catheter
  Other Names: Internal tocodynamometry
  Arms: Intrauterine pressure catheter
Device: External tocodynamometry
  Arms: External tocodynamometry

SUMMARY:
In this study, parturients will be randomized to either internal or external tocodynamometry contractions' follow up. Investigators recruit primiparous, those who try to have vaginal birth after cesarean section and multiparous, who need oxytocin during labor. Primary endpoint is the number of operative labors in each group. Secondary endpoints are the duration of labor, the use of oxytocin and the condition of the newborn.

ELIGIBILITY:
Inclusion Criteria:

* gestational age ≥ 37 weeks
* singleton pregnancy
* a fetus in cephalic position
* normal cardiotocograph in the time of randomization
* cervical ripening < 7 cm
* either 1) primipara, 2) multipara, who needs oxytocin during first stage of labor or 3) parturients with previous cesarean section

Exclusion Criteria:

* parturient with hepatitis or HIV or other significant viral infection
* Acute infections (fever over 37,5, or C-reactive protein over 20) in the time of randomization
* Estimated fetal weight over 4,5 kg
* Suspected fetal abnormality

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1500 (Actual)
Dates: Start 2012-11; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Number of cesarean sections | through study completion, an average of 6 years
Number of operative vaginal deliveries | through study completion, an average of 6 years

SECONDARY OUTCOMES:
Duration of labor | From time of first regular contraction to birth
Newborn admission to the pediatric care unit | 3 days after birth
The use of Oxytocin during labor | From beginning of the use of oxytocin to the birth
Apgar scores | 10 min after birth
Ph of umbilical artery | immediately after birth

CONTACTS AND LOCATIONS:
Overall Officials: Tuija Hautakangas, MD, Principal Investigator — Central Finland Central Hospital, Tampere University
Locations (2):
- Finland (2):
  - Cetral Finland Central Hospital, Jyväskylä, Central Finland
  - Tampere University Hospital, Tampere, Pirkanmaa

IPD SHARING:
Plan to Share IPD: No